CLINICAL TRIAL: NCT00661869
Title: Outcome Evaluation of Solutions for Wellness and Team Solutions Program in Patients With Severe Mental Illness
Acronym: Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Jean-Pierre Lindenmayer, Manhattan Psychiatric Center & NYU School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05I/C51-3
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Wellness Group (Active Comparator)
  Interventions: Other: Wellness Program

INTERVENTIONS:
Other: Wellness Program — 36 weeks of educational and supportive interventions

SUMMARY:
Obesity is increasing at an alarming rate in patients with schizophrenia, possibly in association with the increased use of atypical antipsychotics. In order to address the weight and metabolic syndrome issues, Manhattan Psychiatric Center (MPC) has implemented the Solutions for Wellness and Team Solutions Program. This program is designed to create a supportive, educational and monitoring environment to stabilize both the psychiatric and medical conditions and to prepare patients for independent management of their psychiatric and physical health condition in the community.

DETAILED DESCRIPTION:
The present program is divided into five detailed segments with three progressive levels, that provide a manualized lesson-by-lesson curriculum for implementation on the treatment mall.

* Medication Education
* Symptom recognition and management
* Living Healthy
* Interpersonal Skills
* Discharge Preparation

The program comprised of detailed instructor and patient manuals, specific curriculums and pre- and post-tests to determine acquisition of the learned materials. All modules are imbedded in weekly small group sessions.

* Each of the 5 modules are discussed in groups in weekly morning or afternoon session, Monday through Friday.
* Each module is divided into three 12-week periods for a total of 36 sessions.
* Upon completing 12 weeks at Level 1, each patient moves to Level 2 and then Level 3 for 12 weeks each.
* Each group has two trained instructors.
* Number of patients per group: ≤ 15.
* Sessions are interspersed within the patient's regular treatment mall classes

ELIGIBILITY:
Inclusion Criteria:

1. Are at lease 18 years of age; ≤ 65 years.
2. Are male or female
3. Are currently hospitalized at Manhattan Psychiatric Center and attend daily treatment mall programs.
4. Are fluent in the language of the investigator, and study staff (including testing administrators, group leaders and supervisors)
5. Have a documented current psychiatric diagnosis as obtained from patient's medical charts and recorded by a qualified psychiatrist.
6. Recently admitted patients will be included if their clinical state permits it.

Exclusion Criteria:

1. Are > 65 years of age;
2. Are currently enrolled in the Intensive Psychiatric Services (IPS) program at Manhattan Psychiatric Center;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pre and post-test knowledge assessments attained from each module | 36 weeks
Change in weight, abdominal girth, blood pressure, metabolic markers (Glucose , Insulin, C-peptide, Glycohemoglobin, total cholesterol, total triglycerides, HDL and LDL, leptin, and free fatty acid (FFA)) | 36 weeks

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, M.D., Principal Investigator — New York University School of Medicine & Manhattan Psychaitric Center
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

REFERENCES:
- [Background] Menza M, Vreeland B, Minsky S, Gara M, Radler DR, Sakowitz M. Managing atypical antipsychotic-associated weight gain: 12-month data on a multimodal weight control program. J Clin Psychiatry. 2004 Apr;65(4):471-7. PMID 15119908
- [Background] Lindenmayer JP, Czobor P, Volavka J, Citrome L, Sheitman B, McEvoy JP, Cooper TB, Chakos M, Lieberman JA. Changes in glucose and cholesterol levels in patients with schizophrenia treated with typical or atypical antipsychotics. Am J Psychiatry. 2003 Feb;160(2):290-6. doi: 10.1176/appi.ajp.160.2.290. PMID 12562575
- See also: The Partners for Excellence in Psychiatry (PEP): Neuroscience Treatment Team Partner (NTTP) and Complete Wellness National Training and Consultation Program — http://130.219.250.123/pepweb/aboutus/index.htm